CLINICAL TRIAL: NCT05177549
Title: Evaluation of Anterior Tibial Translation of the Knee in Healthy Women, at Two Times of the Menstrual Cycle, on Hormonal Contraceptives or Not (FLEX)
Acronym: FLEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-AOI-01
Record Dates: First submitted 2021-11-16; First posted 2022-01-04 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Ligament; Laxity
Keywords: hormonal impregnation
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- on estrogen-progestin contraception (Experimental)
  Interventions: Other: Bilateral knee examination with Lachmeter®
- under micro-progestational contraception (Experimental)
  Interventions: Other: Bilateral knee examination with Lachmeter®
- without hormonal contraception (Experimental)
  Interventions: Other: Bilateral knee examination with Lachmeter®

INTERVENTIONS:
Other: Bilateral knee examination with Lachmeter® — Bilateral knee examination with Lachmeter®. Examination repeated 3 times on each knee

SUMMARY:
Women's participation in sports at all levels has been increasing in recent decades. Many individual and team sports are at risk of anterior cruciate ligament (ACL) injury. This injury leads to a permanent or long-lasting interruption of sports practice and to significant medical and economic expenses. Women are recognized as being more at risk of anterior cruciate ligament injury with a risk 6 times higher than men. Hyperlaxity is a risk factor for anterior cruciate ligament injury, but the pathophysiological bases are little studied. Hormonal impregnation and certain periods of the menstrual cycle (ovulatory phase) are risk factors for anterior cruciate ligament injury. It therefore seems interesting to investigators to study the influence of hormonal impregnation on ligament laxity. To date no study has investigated such a relationship.

ELIGIBILITY:
Inclusion Criteria:

* Woman between 18 and 40 years old
* No history of surgery of the 2 lower limbs
* No change in contraceptive method in the last 6 months
* Signature of the informed consent
* Affiliation to the social security system
* To be at Day 14 of her menstrual cycle (+/-1 day) (the first day of the cycle (Day1) being considered as the first day of the menstrual period), except for those on micro-progestative contraception not regulated

By inclusion group:

- For women without hormonal contraception: No method of contraception Or a copper intrauterine device Regular cycles of 26 to 33 days

- For women on estrogen-progestin contraception: Correct use of the estrogen-progestin pill according to the MA Or wearing a vaginal ring according to the MA protocol Or wearing a contraceptive skin patch according to the MA protocol Regular cycles of 26 to 33 days

- For women on micro-progestin contraception : Continuous use of the micro-progestogen pill Or wearing a subcutaneous hormonal implant,

Exception: women on micro-progestin contraception who are not regulated:

* They may have an irregular cycle or no cycle to be included
* They can be included on any day if they have no cycle

Exclusion Criteria:

* Pregnancy or breastfeeding in progress
* Hormonal intrauterine device or injectable contraception
* Menopause (defined as no menstruation for one year)
* Surgery: tubal ligation, oophorectomy, adnexectomy, hysterectomy
* History of microcrystalline or infectious pathology localized to the knee
* History of systemic or localized inflammatory joint disease of the knee
* History of fracture, severe sprain or dislocation of the knee joint
* History of osteoarticular or congenital diseases that may lead to laxity (Marfan syndrome, trisomy 21, Ehlers-Danlos syndrome...)
* Sign of hyperlaxity evaluated by a Beighton score higher than 4 (see appendix)
* BMI > 25
* Daily alcohol consumption above the thresholds recommended by Public Health in France (more than 2 glasses per day)
* Woman unable to understand the protocol
* Intense or unusual physical exercise during the last 72 hours (e.g.: marathon, triathlon, competitive cycling race...)
* Woman under guardianship, curatorship or deprived of liberty

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2024-06-08 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
anterior tibial translation of the knee | Day1 (inclusion visit)
  The anterior tibial translation of the knee will be considered as representative of the anterior laxity of the knee of women under hormonal contraception via the Lachman test at 30° measured with a digital arthrometer type Lachmeter® (bilateral examination repeated 3 times on each knee).The degree of laxity will be evaluated thanks to the international classification IKDC:
  * Grade A 0 to 2 mm = normal
  * Grade B 3 to 5 mm = almost normal
  * Grade C 6 to 10 mm = abnormal
  * Grade D > 10 mm = severely abnormal

CONTACTS AND LOCATIONS:
Overall Officials: Christian ROUX, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France